CLINICAL TRIAL: NCT06595004
Title: A Randomized, Double-blind, Active-controlled, Non-inferiority, Multicenter Phase III Study to Evaluate the Efficacy and Safety of HCP1004 as Compared to RLD2401 in Chronic Low-Back Pain Patients
Brief Title: A Study to Evaluate the Efficacy and Safety of HCP1004 in Chronic Low-Back Pain Patients
Acronym: LBP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-NEON-301
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental 1 (Experimental): Take HCP1004 twice daily for 12 weeks orally.
  Interventions: Drug: HCP1004
- Active Comparator (Active Comparator): Take RLD2401 twice daily for 12 weeks orally.
  Interventions: Drug: RLD2401

INTERVENTIONS:
Drug: HCP1004 — Test Drug
  Arms: Experimental 1
Drug: RLD2401 — Reference drug
  Arms: Active Comparator

SUMMARY:
A Randomized, Double-blind, Active-controlled, Non-inferiority, Multicenter Phase III Study to Evaluate the Efficacy and Safety of HCP1004 as compared to RLD2401 in Chronic Low-Back Pain Patients

ELIGIBILITY:
Inclusion Criteria:

1. Chronic low back pain ≥3 months in duration
2. Quebec Task Force in Spinal Disorders class 1 or 2
3. Male or female ≥ 19 years of age with following criteria:

   * ≥ 50 years
   * 19~ 49 years with history of gastric or duodenal ulcers within the past 5 years
   * Low back pain disease condition expected to require daily NSAIDs therapy for at least 12 weeks
4. VAS ≥ 40 (at Visit 2) (If there are any treatment history to affect the efficacy evaluation of low back pain, VAS after washout period have to meet the criteria; 20% over baseline VAS or change from baseline VAS ≥10)

Exclusion Criteria:

1. Diagnosed with certain serious diseases that may be secondary causes of Low back pain (e.g., tumors, infectious diseases, gout, etc.)
2. Clinically significant neurological disease or low back pain due to trauma (e.g. spinal fracture) within the past 6 months
3. Invasive procedures (using corticosteroids) in the lumbar region within the past 3 months or surgical intervention within the past 6 months or need to such interventions during the study
4. History of non-drug treatment of the lumbar region (e.g., physical therapy) for the purpose of alleviating low back pain within 7 days prior to the screening visit.
5. Active gastritis, inflammatory bowel syndrome, peptic ulcer or any history of gastrointestinal bleeding duodenal ulceration within the past 3 months
6. Patients with history of platelet-related disease or bleeding disorder within the past 6 months or who are taking anti-coagulants
7. Patients with ischemic heart disease or severe cerebrovascular disease within the past 6 months
8. Bronchial asthma or Uncontrolled Diabete Mellitus or Hypertension
9. Use of peptic ulcer treatment (H2-blockers, PPI, PCAB series or Misoprostol), psychotropic drugs, narcotic analgesics or systemic corticosteroids within past 4 weeks
10. Severe renal dysfunction (Creatinine clearance ≥ 30mL/min ) or Severe liver dysfunction (AST or AST ≥ 3 x UNL)
11. History of malignant tumors within past 5 years
12. Positive to pregnancy test, nursing mother, intention on pregnancy
13. Considered by investigator as not appropriate to participate in the study with other reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in VAS | 4 weeks

SECONDARY OUTCOMES:
Change from baseline in VAS(Visual Analog Scale) | 8 weeks, 12 weeks
Change from baseline in ODI(Oswestry Disability Index) Score | 4 weeks, 8 weeks, 12 weeks
Change from baseline in EQ-5D Score | 4 weeks, 8 weeks, 12 weeks
Change from baseline in GSRS(Gastrointestinal Symptom-Rating Scale) Score | 4 weeks, 8 weeks, 12 weeks
Usage of rescue medicine | 4 weeks, 8 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Seoul Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No